CLINICAL TRIAL: NCT01531179
Title: Role Of Lactobacillus Reuteri in Preventing Necrotizing Enterocolitis in Very Low Birth Weight Infants
Brief Title: Lactobacillus Reuteri for Prevention of Necrotizing Enterocolitis in Very Low-birth Weight Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Principal Investigator, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZTB6303
Record Dates: First submitted 2012-02-04; First posted 2012-02-10 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-02

CONDITIONS: Necrotizing Enterocolitis; Very Low Birth Weight Infants
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus reuteri (Experimental): Lactobacillus reuteri 100 million CFU/day for 3 months
  Interventions: Drug: Lactobacillus reuteri
- Control (Placebo Comparator): Placebo for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus reuteri — Lactobacillus reuteri 100 million CFU/day for 3 months
  Other Names: BioGaia
  Arms: Lactobacillus reuteri
Drug: Placebo — Placebo for 3 months
  Arms: Control

SUMMARY:
Probiotics are favorable microorganisms that regulate the flora of the gastrointestinal system and stimulate the immune system. Necrotizing enterocolitis incidence is 10-25% in newborn infants whose birth weights are < 1500 g. Although bifidobacterium and other lactobacilli spp. have been used to reduce the incidence of necrotizing enterocolitis in clinical trials, Lactobacillus reuteri has not been used in the prevention of necrotizing enterocolitis in very low birth weight infants yet. The objective of this study is to evaluate the efficacy of orally administered Lactobacillus reuteri in reducing the incidence and severity of necrotizing enterocolitis in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants < 1500 gr
* Gestational age < 32 weeks

Exclusion Criteria:

* Genetic anomalies
* Short bowel syndrome
* Not willing to participate
* Allergy to Lactobacillus reuteri components

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effect of Lactobacillus reuteri on necrotizing enterocolitis in VLBW infants | up to 6 months
  NEC diagnosis will make modified Bell's criteria. Grade 1A will not include in NEC group.

SECONDARY OUTCOMES:
Effect of Lactobacillus reuteri on culture proved sepsis | up to 6 months
  Patients with culture positivity will accept as proven sepsis.
Effect of Lactobacillus reuteri on weight gain | up to 6 months
  The infants will be weight daily on scales that will calibrated weekly.
Effect of Lactobacillus reuteri on length of hospital stay | up to 6 months
  Specified length of hospital stay as days

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yekta Oncel, MD, Principal Investigator — Neonatology
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Neonatology Unit, Ankara, Turkey, Turkey (Türkiye)

REFERENCES:
- [Derived] Oncel MY, Sari FN, Arayici S, Guzoglu N, Erdeve O, Uras N, Oguz SS, Dilmen U. Lactobacillus Reuteri for the prevention of necrotising enterocolitis in very low birthweight infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F110-5. doi: 10.1136/archdischild-2013-304745. Epub 2013 Dec 5. PMID 24309022
- See also: Lactobacillus reuteri — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=L040030000&QV1=LACTOBACILLUS+REUTERI